CLINICAL TRIAL: NCT00980993
Title: Pilot Study on the Quantification of Respiratory-induced Prostate Motion During Radiation Therapy Using Continuous Real-time Tracking
Brief Title: Quantification of Respiratory-induced Prostate Motion
Status: Withdrawn | Type: Observational
Why Stopped: Lack of enrollment.
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Other Study IDs: OHSU IRB00005606
Record Dates: First submitted 2009-09-19; First posted 2009-09-21 (Estimated); Last update posted 2019-11-04 (Actual); Status verified 2019-10

CONDITIONS: Prostate Cancer
Keywords: Prostate; Motion; Respiration
MeSH Terms: conditions — Prostatic Neoplasms; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patient anatomy and position during the course of radiation therapy can vary from those used for treatment planning; a function of patient movement, uncertainty in positioning system, and organ motion. Traditionally, treatment margins are designed to compensate for interfraction prostate setup variability. This approach has the potential to lower the overall effectiveness of treatment because the prostate gland is a continuously moving target whose motion cannot be accurately accounted for solely on the basis of interfraction movement. More recently, the dosimetric relevance of intra-fraction prostate motion has been recognized, and may be compensated for by continuous real-time adaptive radiation therapy afforded by the Calypso 4D Localization System™. In the current study, the investigators propose to characterize intrafraction prostate motion. The investigators hypothesize that intrafraction prostate motion is correlated with respiratory motion.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed stage I-III adenocarcinoma of the prostate gland
* Age > 18 years. Males of all races and ethnic groups
* Scheduled to receive radiation for definitive therapy
* Three (3) electromagnetic transponders implanted into prostate gland

Exclusion Criteria:

* Does not satisfy inclusion criteria

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Localized prostate cancer patients undergoing intensity-modulated radiation therapy.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2013-09 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Motion amplitude | Continuously during radiation administration (generally 8 to 15 minutes in duration)
  Measured at frequency of 10Hz

CONTACTS AND LOCATIONS:
Overall Officials: James A. Tanyi, Ph.D., Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

REFERENCES:
- See also: Department of Radiation Medicine, Oregon Health and Science University — http://www.ohsu.edu/radmedicine